CLINICAL TRIAL: NCT04519892
Title: A Pilot Study of the Effect of Personalized Depression Risk Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, JianLi Wang, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: pilot#1
Record Dates: First submitted 2020-08-07; First posted 2020-08-20 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Depression; Psychological Distress
Keywords: risk communication; self-help; mental health service use
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with two arms. After screening and baseline assessment, participants will be randomized into: (1) Control group: Receiving PDRC only, and (2) Intervention group: Receiving PDRC + coach guidance. The trial was designed to compare the costs and effectiveness between the groups to inform future implementation. The randomization will be conducted in males and females separately because the MVRPs are sex-specific and the thresholds of high-risk differ by sex. Participants will be assessed at baseline and 3-month.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Over the study period, investigators will be blinded to participants' group status. The survey firm interviewers who conduct randomization, will not be involved in follow-up interviews. The interviewers who conduct the follow-up interviews in Ottawa will not have access to participants' group status. The coaches will not be involved in follow-up assessments. Given our description of study objectives, some participants may know their group status. Therefore, it is possible that some participants in the control group may try to find more information about the PDRC. At the follow-up assessments, participants will be asked if they have used any risk prediction tools over the study period. At the follow-up assessments, if participants develop a MDE, they will be encouraged to contact their family doctors and information about local mental health resources will be provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving PDRC and coach guidance (Experimental): Intervention group: Receiving PDRC + coach guidance.
  Interventions: Other: PDRC; Other: Coach guidance
- Receiving PDRC without coach guidance (Active Comparator): Control group: Receiving PDRC only.
  Interventions: Other: PDRC

INTERVENTIONS:
Other: PDRC — Personalized depression risk communication.
Other: Coach guidance — Coaching service to guide the understanding of PDRC and answer questions.
  Arms: Receiving PDRC and coach guidance

SUMMARY:
Depression is a highly prevalent and disabling mental health problem. It is associated with significant morbidity and mortality and it has a significant economic impact. Effective and feasible strategies aimed at the population-level to reduce the risk of onset are urgently needed to manage this ubiquitous condition. Developed from research in the fields of epidemiology, mental health, and implementation science, the proposed intervention provides individualized information designed to trigger actions that can reduce the risk of MDE. Specifically, and as the first step, the investigators developed the first sex-specific multivariable risk predictive algorithms (MVRPs) for MDE using data from over 10,000 Canadians. This innovative early work shows that the risk of onset of MDE can be quantified in the same way as can other physical disorders such as cardiovascular diseases and cancer. Knowing the individualized risk estimated by the MVRPs may serve as a trigger to empower people to actively engage in effective self-help actions. Self-help strategies are commonly used to deal with depression and promoting effective self-help strategies to the public as an early intervention strategy has been recommended as one way to reduce the large disease burden of depression. Subsequently, the investigators conducted a randomized controlled trial (RCT) and found that providing individualized depression risk causes no psychological harm in participants. These studies have laid the required foundation for communicating individualized risk information to a broad population as a first step towards effecting changes in self-help and help-seeking behaviours and reducing the risk of MDE onset.

Using the MVRPs as the foundation and working with future users, the investigators developed a personalized depression risk communication tool (PDRC) for sharing information about individualized depression risk, risk profile (risk factors present), potential risk reduction, and self-help strategies. At this stage of our research program, the investigators need to answer the question: Does the PDRC lead to positive changes in self-help and help-seeking behaviours? Prior to a large scale RCT, the investigators proposed to conduct a pilot study to gain preliminary understanding about the effect of PDRC on self-help and help-seeking behaviors. The results will inform the design of a large RCT.

DETAILED DESCRIPTION:
Depression is a highly prevalent and disabling mental health problem. It is associated with significant morbidity and mortality and it has a significant economic impact. Effective and feasible strategies aimed at the population-level to reduce the risk of onset are urgently needed to manage this ubiquitous condition. Developed from research in the fields of epidemiology, mental health, and implementation science, the proposed intervention provides individualized information designed to trigger actions that can reduce the risk of MDE. Specifically, and as the first step, the investigators developed the first sex-specific multivariable risk predictive algorithms (MVRPs) for MDE using data from over 10,000 Canadians. This innovative early work shows that the risk of onset of MDE can be quantified in the same way as can other physical disorders such as cardiovascular diseases and cancer. Knowing the individualized risk estimated by the MVRPs may serve as a trigger to empower people to actively engage in effective self-help actions. Self-help strategies are commonly used to deal with depression and promoting effective self-help strategies to the public as an early intervention strategy has been recommended as one way to reduce the large disease burden of depression. Subsequently, the investigators conducted a randomized controlled trial (RCT) and found that providing individualized depression risk causes no psychological harm in participants. Using the MVRPs as the foundation and working with future users, the investigators developed a personalized depression risk communication tool (PDRC) for sharing information about individualized depression risk, risk profile (risk factors present), potential risk reduction, and self-help strategies.

Risk communication is the open two way exchange of information and opinions about harms and benefits, with the aim of improving the understanding of risk and of promoting better decisions about clinical management. Risk communication goes beyond simply sharing information about the probability of developing a problem (i.e., individualized risk); it also shares possible actions to be taken. The notable clinical guidelines for coronary heart disease (CHD) and the Institute of Medicine report recommend that baseline risk should be estimated; individuals should know their personal risk; and high-quality risk communication tools should be developed.

The existing literature reveals that effective risk communication often includes multiple components: (1) Individualized risk information presented as an absolute risk, as opposed to a relative risk. The risk information may also list the individual's risk factors. (2) Appropriate format of presentation (e.g., graphic, visual). The format of presentation can influence the degree to which individuals perceive their risk and will affect behavioural change. (3) Presentation of risk reduction. A review of evidence recommends that information on risk reduction should be presented using absolute risk reduction. Presenting the risk reduction of behavioural change to the individual is the most commonly used behavioural change technique in the literature. (4) Framing. Describing the consequences of performing or not performing an action, presented as a gain versus a loss,18 and (5) Decision aids to help consumers participate in decisions by providing clear evidence based information on available choices. Personalized risk communication tools with these components are instrumental for making informed decisions regarding the uptake of preventive measures, adhering to risk-reducing therapy, and improving risk perception and health-related behaviours. In mental health, self-help and help-seeking are particularly important for reducing the disease burden of mental disorders. However, changing health-related behaviours to improve mental health and encouraging help-seeking have been very challenging. Based on the theoretical model and the experience of other medical disciplines (to be described below), risk communication may offer a unique opportunity for promoting behaviour change, and if successful, will make a significant contribution to depression prevention.

The principle research question of the proposed study is: Are individuals who are at high risk of having a MDE and who receive the coach-guided PDRC more likely to take self-help actions than those who receive the PDRC without coach guidance? It was hypothesized that high risk people who receive the coach-guided PDRC are more likely to take self-help actions than those receive the PDRC without coach guidance.

The secondary research questions include:

1. What are the impacts of receiving the coach-guided PDRC on psychological distress, depressive symptoms and mental health service use?
2. What are the demographic and clinical factors associated with the behavioural changes?

This is a randomized controlled trial with two arms. After screening and baseline assessment, participants will be randomized into: (1) Control group: Receiving PDRC only, and (2) Intervention group: Receiving PDRC + coach guidance. The trial was designed to compare the costs and effectiveness between the groups to inform future implementation. The randomization will be conducted in males and females separately because the MVRPs are sex-specific and the thresholds of high-risk differ by sex. Participants will be assessed at baseline and 3-month. After each assessment, the following materials will be mailed to participants: (1) a thank-you letter, including the date of the next interview. (2) Self-help strategies34 and a summary of research evidence supporting the effectiveness of the self-help strategies, and (3) a $20 incentive as appreciation for their participation. Participants in the PDRC+coach arm will have access to coach to guide them. Participants in the control group will receive their PDRC only if they are interested.

The recruitment, baseline assessment and randomization will be contracted to a telephone interview firm. The target population of the study are individuals who are at high risk of having a MDE in Canada. Telephone recruitment using the random digit dialing method, screening and data collection are a feasible and economic way for the proposed study. A random sample of landline and cell phone numbers will be selected. When a household is reached, the person who is 18+ years will be assessed for eligibility. If a household has 2+ persons aged 18+ years, one will be randomly selected. The interviewers will explain the study objectives and procedures and answer questions. Oral consent will be obtained before assessment of eligibility.

Screening: Once a potentially eligible participant is identified, the interviewer will confirm the participant's age and administer the Composite International Diagnostic Interview - Major Depression (CIDI) MDE module and the sex-specific MVRPs via telephone. The CIDI is a fully structured diagnostic interview for mental disorders, that is commonly used in community-based mental health surveys, and can be administered by trained lay interviewers. Interviewees who have a MDE at the time of the interview or are below the risk thresholds based on the MVRPs, will be excluded. Individuals with an ongoing MDE will be encouraged to contact their family doctors and information about local mental health resources will be provided. For those who are at low risk, the web site of the MVRPs will be provided so they may monitor their risk in the future.

Baseline assessment: In eligible participants, the interviewer will administer the questionnaire about self-help behaviours, mental health service use, depressive symptoms and quality of life.

Randomization will be carried out in male and in female participants separately. Most survey firms use a survey software built by VOXCO. The tool contains a random number generator which randomly creates a digit when the telephone script reads the function. This randomization approached was used in the IMPACT trial, and the intervention and control groups of the trial were similar in baseline characteristics.

The survey firm will securely transfer encrypted baseline data to the project coordinator on a daily basis. The group assignment data will be transferred in a separate file. The follow-up assessments will be conducted at the PI's telephone interview laboratory at the Institute of Mental Health Research (IMHR). One month before the scheduled follow-up interviews, letters will be sent to participants to remind them of the upcoming interview. After the 3-month interview, group status will be linked with interview data by study ID numbers.

Over the study period, investigators will be blinded to participants' group status. The survey firm interviewers who conduct randomization, will not be involved in follow-up interviews. The interviewers who conduct the follow-up interviews in Ottawa will not have access to participants' group status. The coaches will not be involved in follow-up assessments. Given our description of study objectives, some participants may know their group status. Therefore, it is possible that some participants in the control group may try to find more information about the PDRC. At the follow-up assessments, the investigators will ask if they have used any risk prediction tools over the study period. At the follow-up assessments, if participants develop a MDE, they will be encouraged to contact their family doctors and information about local mental health resources will be provided.

Duration of intervention. The intervention includes delivering the PDRC report via email and coach guidance in its interpretation and planning self-help actions. The PDRC will be sent to the participants within one week after randomization and the coach will initiate contact the following week.

ELIGIBILITY:
Inclusion Criteria:

* no MDE at baseline, and full remission for 2 months for those who had a past MDE (see below the question).
* Aged 18+.
* At high risk of MDE based on the algorithms (predicted risk of 6.5%+ for men and 11.2%+ for women).1
* Agreement to be contacted for follow-up assessments, and
* no language barriers to English or French. The status of remission will be assessed by the question: "In the past 2 months or longer, has your mood been much improved or back to normal AND you DIDN'T have the symptoms?"

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in self-help scores | between baseline and immediate post-intervention
  Self-help behaviors measured by SSUS. The score ranges from 0 to 70 with a higher score indicating more frequent use of self-help.

SECONDARY OUTCOMES:
Non-specific psychological distress | Past 4 weeks
  Psychological distress measured by K10. K10 score ranges from 10 to 50 with a higher score indicating more severe psychological distress.
Depression | Past 2 weeks
  Depressive symptoms measured by PHQ-9. The PHQ-9 score ranges from 0 to 27 with a higher score indicating more depressive symptoms.
Mental health service use | Past 3 months.
  Questions about if in-person or phone contacts were made with health professionals for mental health problems. The same questions used in the Canadian national mental health survey will be adopted. The measurement is not a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jianli Wang, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa Institute of Mental Health Research, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a pilot study to gather information for a large trial.